CLINICAL TRIAL: NCT04126915
Title: Precise Therapy for mCRPC Patients Through Whole Exome Sequencing
Brief Title: Precise Therapy for mCRPC Patients Through Whole Exome Sequencing(PTtWES)
Acronym: PTtWES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yinghao Sun (Other)
Responsible Party: Sponsor-Investigator, Yinghao Sun, MD,Clinical Professor, Changhai Hospital
Organization: Changhai Hospital (Other)
Other Study IDs: mCRPC-WES2019
Record Dates: First submitted 2019-09-24; First posted 2019-10-15 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Castration-Resistant Prostatic Cancer
Keywords: Castration-Resistant Prostatic Cancer; Whole Exome Sequencing
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Biospecimens are metastatic tissues of patients, including bone metastases and metastatic lymph nodes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Whole Exome Sequencing — Whole Exome Sequencing of the patient's primary tumor, metastases

SUMMARY:
Through gene sequencing of the patient's tissue, to figure out the genomic characteristics of patients with advanced disease and guide the treatment of patients

DETAILED DESCRIPTION:
Tumor heterogeneity and tumor clonal evolution cause he diagnosis and treatment difficulties of advanced prostate cancer. Heterogeneity exists in different lesions at the same location of the same tumor, between lesions at different locations, and in the same lesion in different processes of disease progression. Tumor heterogeneity causes different tumor patients to respond differently to different treatments; as patients progress, tumor patients gradually develop clonal evolution, and the original effective treatment will lose the therapeutic effect. And routine imaging examinations and PSA examinations are also difficult to respond to changes in the patient's condition in a timely manner. By Genetic testing of the primary tumor, metastases or blood of the patient, and according to the test result of the patient, the patient's medication treatment can be provided, and the patient's condition change can be monitored. Studies have shown that patients with different mutation types respond differently to the same treatment. Prostate cancer patients with AR-V7 mutations have a poorer response to abiraterone or dextrozamide than patients with prostate cancer without AR-V7 mutation; whereas for solid tumors with MSI-H or dMMR, PD-1 Inhibitors can also bring the desired results to such patients. Therefore, according to the genetic test results of the patient's tumor tissue, early diagnosis can also be given, and the patient's condition change and precise treatment can be predicted.In this study, the investigators hope to obtain the genome characteristics of advanced patients by performing whole exon sequencing on the patient's tissues, and to guide the patients' follow-up treatment through sequencing results, to observe the effects of different treatment methods on patients and find biomarker that predict patient prognosis

ELIGIBILITY:
Inclusion Criteria:

* Expected survival period ≥ half a year;
* Whole body bone scan (ECT) and magnetic resonance imaging (MRI) or PET-CT are evaluated as metastatic castration to resist prostate cancer patients;
* Patients with evaluable and retrievable lesions;
* Patients who voluntarily receive the experimental study protocol after informing the existing treatment plan;

Exclusion Criteria:

* Patients with other malignancies, or in acute infection or other severe infections; immunodeficiency virus (HIV), hepatitis C virus (HCV) and/or syphilis-positive patients;
* Patients who have long-term anticoagulant and anti-platelet aggregation drugs (the anticoagulant is discontinued for less than 1 week);
* At the same time suffering from other serious systemic diseases, the researchers believe that it may interfere with the treatment, evaluation and compliance of this test, including severe respiratory, circulatory, neurological, mental, digestive, endocrine, immune, urinary and other systems. disease;
* The patient that it is inappropriate to participate in this clinical trial

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patient with prostate cancer
Study Population: The enrolled patients were mCRPC patients with measurable and retrievable metastases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-08 (Estimated); Primary Completion 2022-10-08 (Estimated); Study Completion 2024-10-08 (Estimated)

PRIMARY OUTCOMES:
The genetic characteristics of mCRPC patients in China | June 2020
  The genetic characteristics of mCRPC patients in China as Assessed by Gene Sequencing

SECONDARY OUTCOMES:
the possible prognostic therapeutic target | June 2023
  the possible prognostic therapeutic target as Assessed by Gene Sequencing ，by observing the patient's prognosis，including PSA progression and progression in imaging by RECIST Version 1.1
The best method to treat the disease | June 2023
  Compare the effects of different treatments on the prognosis of patients as Assessed by PSA progression and progression in imaging by RECIST Version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: yinghao sun, PHD, Study Chair — Department of Urology，Changhai Hospital of Second Military Medical University

IPD SHARING:
Plan to Share IPD: No